CLINICAL TRIAL: NCT02467764
Title: Definition of a "Score Infectivity" During Reoperation on Total Hip or Knee Prosthesis
Brief Title: "Score Infectivity" During Reoperation on Total Hip or Knee Prosthesis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-20
Record Dates: First submitted 2015-05-14; First posted 2015-06-10 (Estimated); Last update posted 2015-06-10 (Estimated); Status verified 2015-06

CONDITIONS: Osteoarthritis
Keywords: Knee; Knee osteoarthritis; Knee replacement; Hip; Hip osteoarthritis; Hip replacement
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip | interventions — Retrospective Studies

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Retrospective study

SUMMARY:
The hip or knee is a validated treatment of end-stage osteoarthritis, and these interventions commonly make a significant improvement in the quality of life of patients. Infection can occur in 1-5% of cases. Diagnosis is often difficult, but the knowledge of infected or not infected character directly influences the surgical conduct. It is therefore recommended that the positive or negative diagnosis is made in the most reliable way possible, but no single element only allows a low diagnosis. The concomitant use of several clinical, radiological and aggregated into a composite score history could help facilitate this preoperative approach during reoperation on prosthetic joint

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years
* Patients operated in the service in 2014 to care for end-stage hip or knee osteoarthritis by implantation of a total hip or knee prosthesis.

Exclusion Criteria:

* Patients under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients operated in the service in 2014 to care for end-stage hip or knee osteoarthritis by implantation of a total hip or knee prosthesis.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-05 (Estimated); Study Completion 2016-05 (Estimated)

PRIMARY OUTCOMES:
define a composite score on total Hip or Knee Prosthesis | patient's medical data will be collected by health professional for the duration hospital stay, up to 1 year]

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves JENNY, MD, Principal Investigator — University Hospital, Strasbourg, France